CLINICAL TRIAL: NCT02322463
Title: Ethnicity and Analgesic Practice in a Pediatric Emergency Department
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0533-14-RMB-CTIL
Record Dates: First submitted 2014-12-06; First posted 2014-12-23 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Limb Fracture
Keywords: patients who were admitted to the pediatric ED

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arab children (case subjects): Arab patients who were admitted to the pediatric ED due to a limb fracture between 01 January 2011 and 31 October 2014, who were treated with Oxycodone
  Interventions: Drug: Arab children
- Jewish children (controls): Jewish patients who were admitted to the pediatric ED due to a limb fracture between 01 January 2011 and 31 October 2014, who were treated with Oxycodone
  Interventions: Drug: Arab children

INTERVENTIONS:
Drug: Arab children — Treatment with Oxycodone
  Other Names: Arabs

SUMMARY:
Early and appropriate pain management in the emergency department (ED) is an important aspect of child care. Studies in the adult population revealed that ethnicity might be associated with disparities in analgesia and opioid treatment in ED patients suffering from limb fractures. The investigators aim to explore if ethnicity has an influence on analgesic practice in the pediatric ED. The objective of this study is to determine whether minority population Arab children with orthopedic injuries are less likely than Jewish children to receive oxycodone for limb fracture.

DETAILED DESCRIPTION:
Early and appropriate pain management in the emergency department (ED) is an important aspect of child care. Studies in the adult population revealed that ethnicity might be associated with disparities in analgesia and opioid treatment in ED patients suffering from limb fractures. The investigators aim to explore if ethnicity has an influence on analgesic practice in the pediatric ED. The objective of this study is to determine whether minority population Arab children with orthopedic injuries are less likely than Jewish children to receive oxycodone for limb fracture .

ELIGIBILITY:
Inclusion Criteria:

-Any patient with a limb fracture

Exclusion Criteria:

* Multi trauma patients
* Patients with unidentified ethnicity

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients who were admitted to the pediatric ED due to a limb fracture between 01 January 2011 and 31 October 2014
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Rate of oxycodone treatment by the nursing staff | At triage up to 1 hour after admission at the recpetion desk

CONTACTS AND LOCATIONS:
Overall Officials: ITAI Shavit, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

REFERENCES:
- [Derived] Shavit I, Brumer E, Shavit D, Eidelman M, Steiner IP, Steinberg C. Emergency Department Pain Management in Pediatric Patients With Fracture or Dislocation in a Bi-Ethnic Population. Ann Emerg Med. 2016 Jan;67(1):9-14.e1. doi: 10.1016/j.annemergmed.2015.07.497. Epub 2015 Sep 3. PMID 26343348